CLINICAL TRIAL: NCT05872620
Title: A Phase 3, Randomized, Double-Blind Study to Investigate the Efficacy and Safety of Once-Daily Oral LY3502970 Compared With Placebo in Adult Participants With Obesity or Overweight and Type 2 Diabetes (ATTAIN-2)
Brief Title: A Study of Orforglipron in Adult Participants With Obesity or Overweight and Type 2 Diabetes
Acronym: ATTAIN-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18560; J2A-MC-GZGQ (Other: Eli Lilly and Company); 2022-502837-24-00 (Other: Eli Lilly and Company); U1111-1289-8799 (Other: UTN Number)
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Overweight; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2 | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Orforglipron Dose 1 (Experimental): Participants will receive orforglipron administered orally.
  Interventions: Drug: Orforglipron
- Orforglipron Dose 2 (Experimental): Participants will receive orforglipron administered orally.
  Interventions: Drug: Orforglipron
- Orforglipron Dose 3 (Experimental): Participants will receive orforglipron administered orally.
  Interventions: Drug: Orforglipron
- Placebo (Placebo Comparator): Participants will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: LY3502970
  Arms: Orforglipron Dose 1; Orforglipron Dose 2; Orforglipron Dose 3
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
This study will investigate the safety and efficacy of once daily oral treatment with orforglipron compared with placebo on body weight in adult participants with obesity or overweight and type 2 diabetes. The study will last about 77 weeks and may include up to 22 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) ≥27.0 kilogram/square meter (kg/m²).
* Have a history of at least 1 self-reported unsuccessful dietary effort to lose body weight.
* Have a diagnosis of Type 2 Diabetes (T2D), with HbA1c ≥7% (≥53 mmol/mol) to ≤10% (86 mmol/mol) and are on stable treatment for T2D for at least 90 days prior to screening, consisting of:

  * either diet/exercise alone or
  * up to 3 oral antihyperglycemic medications (excluding dipeptidyl peptidase IV inhibitors (DPP-4i) or glucagon-like peptide-1 (GLP-1) receptor agonists (RA).

Exclusion Criteria:

* Have Type 1 Diabetes (T1D), history of ketoacidosis or hyperosmolar state/coma, or any other types of diabetes except T2D.
* Have a self-reported change in body weight >5 kg (11 pounds) within 90 days prior to screening.
* Are currently receiving or planning to receive treatment for diabetic retinopathy and/or macular edema (for example, laster photocoagulation or intravitreal injections of anti-vascular endothelial growth factor inhibitors).
* Have family (first-degree relative) or personal history of medullary thyroid cancer (MTC) or multiple endocrine neoplasia 2 (MEN2) syndrome.
* Have had a history of chronic or acute pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1613 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Mean Percent Change from Baseline in Body Weight | Baseline, Week 72

SECONDARY OUTCOMES:
Mean Change from Baseline in Waist Circumference | Baseline, Week 72
Mean Change from Baseline in Hemoglobin A1c (HbA1c) % | Baseline, Week 72
Mean Change from Baseline in Fasting Glucose | Baseline, Week 72
Mean Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 72
Mean Change from Baseline in Fasting Triglycerides | Baseline, Week 72
Mean Percent Change from Baseline in Fasting non-High-Density Lipoprotein (HDL) Cholesterol | Baseline, Week 72
Mean Percent Change from Baseline in Fasting Insulin | Baseline, Week 72
Mean Change from Baseline in Diastolic Blood Pressure (DBP) | Baseline, Week 72
Mean Change from Baseline in Short Form 36 Version 2 Health Survey Acute Form (SF-36v2) Domain Scores | Baseline, Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (136):
- United States (37):
  - Cahaba Research - Pelham, Pelham, Alabama
  - Novak Clinical Research - Tucson - North La Cholla Boulevard, Tucson, Arizona
  - Yuma Clinical Trials, Yuma, Arizona
  - AMCR Institute, Escondido, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Velocity Clinical Research, Westlake, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - University Clinical Investigators, Inc., Tustin, California
  - Encore Medical Research, Hollywood, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - South Florida Clinical Research Institute, Margate, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Balanced Life Health Care Solutions/SKYCRNG, Lawrenceville, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Pacific Diabetes & Endocrine Center, Honolulu, Hawaii
  - Solaris Clinical Research, Meridian, Idaho
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - IMA Clinical Research, Albuquerque, New Mexico
  - Albany Medical College, Division of Community Endocrinology, Albany, New York
  - Albany Stratton VA Medical Center, Albany, New York
  - NYC Research INC, Long Island City, New York
  - Accellacare - Raleigh, Raleigh, North Carolina
  - Summit Headlands, Portland, Oregon
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Soma Clinical Trials, Denison, Texas
  - Epic Medical Research - DeSoto, DeSoto, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Diabetes and Glandular Disease Center, San Antonio, Texas
  - VIP Trials, San Antonio, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Universal Research Group, Tacoma, Washington
- Argentina (11):
  - Mautalen Salud e Investigación, Buenos Aires, Buenos Aires F.D.
  - CEMEDIAB, C.a.b.a., Ciudad Aut
  - Instituto Centenario, CABA, Ciudad Autónoma de Buenos Aire
  - Instituto de Investigaciones Clinicas Rosario, Rosario, Santa Fe Province
  - Instituto Médico Fundación Grupo Colaborativo Rosario Investigación y Prevención Medica, Rosario, Santa Fe Province
  - Sanatorio San Martin, Venado Tuerto, Santa Fe Province
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman, Tucumán Province
  - CONEXA Investigacion Clinica S.A., Buenos Aires
  - Centro Diabetológico Dr. Waitman, Córdoba
  - Clínica Universitaria Reina Fabiola, Córdoba
  - Centro de Diagnóstico y Rehabilitación (CEDIR), Santa Fe
- Australia (11):
  - Emeritus Research, Botany, New South Wales
  - The AIM Centre / Hunter Diabetes Centre, Merewether, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Core Research Group, Brisbane, Queensland
  - Logan Hospital, Meadowbrook, Queensland
  - Southern Adelaide Diabetes & Endocrine Services, Oaklands Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Emeritus Research, Camberwell, Victoria
  - Austin Health - Repatriation Hospital, Heidelberg West, Victoria
  - Baker IDI Heart and Diabetes Institute - Melbourne, Melbourne, Victoria
  - Advara HeartCare Joondalup, Joondalup, Western Australia
- Brazil (8):
  - Centro de Pesquisa Clinica do Brasil, Brasília, Federal District
  - Cendi - Endocrinologia e Diabetes, Goiânia, Goiás
  - Instituto Lóbus, Volta Redonda, Rio de Janeiro
  - Instituto Méderi de Pesquisa e Saúde, Passo Fundo, Rio Grande do Sul
  - Instituto de Pesquisa clinica de Campinas, Campinas, São Paulo
  - Centro de Pesquisa Clínica de Marília - CPCLIM, Marília, São Paulo
  - Pesquisare Saude, Santo André, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
- China (18):
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - ShenZhen People's Hospital, Shenzhen, Guangdong
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Jiangsu Province Official Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nantong First People's Hospital, Nantong, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Dalian Municipal Central Hospital Affiliated of Dalian Medical University, Dalian, Liaoning
  - Jinan Central Hospital, Jinan, Shandong
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Zhu Xianyi Memorial Hospital, Tianjin, Tianjin Municipality
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
- Czechia (12):
  - Milan Kvapil s.r.o., Diabetologicka ambulance Pribram, Příbram, Central Bohemia
  - MUDr. Alena Vachova, České Budějovice, Jihočeský kraj
  - MUDr. Tomas Edelsberger, Krnov, Moravskosl
  - Diahelp s.r.o, Pardubice V, Pardubice
  - Dialine - Interni a diabetologicka ambulance, Pilsen, Plzeň-město
  - Diabet2 s.r.o., diabetologicka a interni ambulance, Prague, Praha 1
  - Milan Kvapil s.r.o., Diabetologicka ambulance, Prague, Praha 4
  - ResTrial s.r.o., Prague, Praha 8
  - MUDr. Sabina Palova, Jílové u Prahy, Praha-západ
  - Nemocnice Cesky Krumlov, Český Krumlov
  - Endokrinologie MUDr. Rehorkova s.r.o., Hradec Králové
  - MUDr. Jitka Zemanová - diabetologie a interna s.r.o., Pilsen
- Germany (15):
  - CDG Studienambulanz Hartard, München, Bavaria
  - Gemeinschaftspraxis Dr. med. Josef und Wilma Großkopf, Wallerfing, Bavaria
  - Ceda-Research, Pohlheim, Hesse
  - Institut für Diabetesforschung GmbH Münster, Münster, Nordrhein-
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - InnoDiab Forschung Gmbh, Essen, North Rhine-Westphalia
  - Medizentrum Essen Borbeck, Essen, North Rhine-Westphalia
  - AmBeNet GmbH, Leipzig, Saxony
  - Arztpraxis Christine Kosch Pirna, Pirna, Saxony
  - Hausarzt- und Diabetologische Schwerpunktpraxis Hohenmölsen - Weiβenfels, Hohenmölsen, Saxony-Anhalt
  - SMO.MD GmbH, Magdeburg, Saxony-Anhalt
  - Universität zu Lübeck - Institut für Endokrinologie und Diabetes, Lübeck, Schleswig-Holstein
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Diabetes Zentrum Dr. Tews, Gelnhausen
  - Diabetes Zentrum Wilhelmsburg, Hamburg
- Greece (7):
  - Athens Medical Center, Athens, Attikí
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki, Kentrikí Makedonía
  - Euromedica General Clinic of Thessaloniki, Thessaloniki, Thessaloníki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki, Thessaloníki
  - Thermi Clinic, Thessaloniki, Thessaloníki
  - University General Hospital of Larissa, Larissa, Thessalía
  - 424 Military General Training Hospital, Thessaloniki
- India (9):
  - Medstar Speciality Hospital, Bangalore, Karnataka
  - Karnataka Institute of Medical Sciences, Hubli, Karnataka
  - TOTALL Diabetes Hormone Institute, Indore, Madhya Pradesh
  - Topiwala National Medical College & B. Y. L. Nair Charitable Hospital, Mumbai, Maharashtra
  - BSES MG Hospital, Mumbai, Maharashtra
  - All India Institute of Medical Sciences (AIIMS) - Nagpur, Nagpur, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Arthur Asirvatham Hospital, Madurai, Tamil Nadu
  - Kumudini Devi Diabetes Research Center, Hyderabad, Telangana
- Puerto Rico (2):
  - Advanced Clinical Research, LLC, Bayamón, PR
  - Isis Clinical Research Center, Guaynabo, PR
- South Korea (6):
  - Yonsei University-Wonju Severance Christian Hospital, Wŏnju, Kang-won-do
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Yeungnam Univeristy Medical Center, Gyeongsan-si, Kyǒngsangbuk-do
  - Korea University Anam Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Kyung Hee University Hospital at Gangdong, Seoul, Seoul-teukbyeolsi [Seoul]

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Time Frame:
  Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Horn DB, Ryan DH, Kis SG, Alves B, Mu Y, Kim SG, Aberle J, Bain SC, Allen S, Sarker E, Wu Q, Stefanski A, Jouravskaya I; ATTAIN-2 Trial Investigators. Orforglipron, an oral small-molecule GLP-1 receptor agonist, for the treatment of obesity in people with type 2 diabetes (ATTAIN-2): a phase 3, double-blind, randomised, multicentre, placebo-controlled trial. Lancet. 2026 Dec 20;406(10522):2927-2944. doi: 10.1016/S0140-6736(25)02165-8. Epub 2025 Nov 20. PMID 41275875
- See also: A Study of Orforglipron in Adult Participants With Obesity or Overweight and Type 2 Diabetes (ATTAIN-2) — https://trials.lilly.com/en-US/trial/404300